CLINICAL TRIAL: NCT05428748
Title: An Open-label, Parallel and Randomized Trial to Assess the Safety and Tolerability of a Novel Hydration Drink in Healthy Volunteers
Brief Title: Clinical Trial to Evaluate Safety and Tolerability of a Novel Hydration Drink in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liquid I.V. (Other)
Collaborators: University of Memphis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SOW5
Record Dates: First submitted 2022-06-15; First posted 2022-06-23 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Tolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1S (Experimental): Participants will consume 1 serving/day of the test product for 28 days.
  Interventions: Other: 1 serving of test product
- 2S (Experimental): Participants will consume 2 servings/day of the test product for 28 days
  Interventions: Other: 2 servings of test product
- 3S (Experimental): Participants will consume 3 servings/day of the test product for 28 days
  Interventions: Other: 3 servings of test product
- Placebo (Placebo Comparator): Participants will consume 1 serving/day of the placebo for 28 days
  Interventions: Other: Placebo

INTERVENTIONS:
Other: 1 serving of test product — Participants will consume 1 serving/day of the test product for 28 days
  Arms: 1S
Other: 2 servings of test product — Participants will consume 2 servings/day of the test product for 28 days
  Arms: 2S
Other: 3 servings of test product — Participants will consume 3 servings/day of the test product for 28 days
  Arms: 3S
Other: Placebo — Participants will consume 1 serving/day of the placebo for 28 days
  Arms: Placebo

SUMMARY:
This clinical trial design aims to evaluate the safety and tolerability of a novel hydration drink in health volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals who are between 18 - 35 years of age. Have a body mass index (BMI) range of 18.0 - 24.9 kg/m2. Willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, be able to understand and read the questionnaires, and carry out all study-related procedures

Exclusion Criteria:

* Participant has a positive medical history of heart disease/cardiovascular disease, uncontrolled hypertension (140/90 or greater mmHg), kidney disease (dialysis or renal failure), hepatic impairment or disease, or Type I or Type II diabetes. Participant has a positive medical history of unstable thyroid disease, previously diagnosed major affective disorder, psychiatric disorder that required hospitalization in the prior year, immune disorder (i.e., HIV/AIDS), a history of cancer (except localized skin cancer without metastases or in situ cervical cancer within 5 years prior to screening visit. Participant has an abnormality or obstruction of the gastrointestinal tract precluding swallowing (e.g. dysphagia) and digestion (e.g., known intestinal malabsorption, celiac disease, inflammatory bowel disease, chronic pancreatitis, steatorrhea). Individuals who are lactating, pregnant or planning to become pregnant during the study. Have a known sensitivity or allergy to any of the study products. Any condition or abnormality that, in the opinion of the investigator, would compromise the safety of the participant or the quality of the study data. History of alcohol or substance abuse in the 12 months prior to screening. Receipt or use of an investigational product in another research study within 28 days prior to baseline/Visit 2

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Safety of test product | 28 days
  To assess the safety of the test product (TP) via comprehensive metabolic panel, complete blood count, urinalysis, vitals, and observed or reported adverse events.
Tolerability of test product | 28 days
  To assess the tolerability of the test product via participant tolerability questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bloomer, PhD, Principal Investigator — University of Memphis
Locations (1):
- The University of Memphis, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No